CLINICAL TRIAL: NCT06257030
Title: The AMARA (As Much As Reasonably Achievable) Study: Radioembolization of Large Inoperable Liver Tumors
Brief Title: The AMARA (As Much As Reasonably Achievable) Study
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Dr. Konstantinos Katsanos, Associate Professor of Interventional Radiology, University Hospital of Patras
Other Study IDs: 735
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- TARE group: (TARE)Transarterial radioembolization is a transcatheter intra-arterial procedure performed by the interventional radiologist for the treatment of primary and secondary hepatic cancers.
  Interventions: Device: Transarterial Radioembolization

INTERVENTIONS:
Device: Transarterial Radioembolization — (TARE)Transarterial radioembolization is a transcatheter intra-arterial procedure performed by the interventional radiologist for the treatment of primary and secondary hepatic cancers.

SUMMARY:
Subjects with large inoperable liver tumors defined as at least 1 lesion larger than 5cm in maximum diameter. For the purposes of the present study, we define the AMARA principle in intensified regional TARE as a planned irradiated tumor dose >200Gy by the partition model. The purpose of the study is to evaluate the safety and efficacy of Y90 high dose radioembolization for the management of large inoperable liver tumors. In addition, to correlate the safety and efficacy with the post-treatment dosimetry analysis (by MIM Software Inc) based on 90Y-PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yr
* Both sexes eligible for study
* Patients with primary or secondary liver tumors
* Liver dominant disease
* At least one lesion greater than 5.0 cm in maximum diameter
* Life-expectancy > 3 months
* FLR >40% or greater than 500mls
* Must be able to tolerate pre-treatment CT scan , DSA and 99mTc-MAA infusion and imaging with SPECT/CT scan
* Able to schedule and tolerate post-treatment Y90 PET/CT imaging
* Able to tolerate follow-up imaging with dynamic contrast CT liver phase or MRI with liver specific contrast at 3mo, 6mo, 9mo, 1yr, 2.0 yr, and 3.0 years.

Exclusion Criteria:

* Child Pugh > B
* Bilirubin >2 mg/dl
* Albumin<3.0
* Central portal invasion
* Multi-focal bilobar disease
* Disseminated extrahepatic disease
* Lung shunt >20% or a estimated Lung dose > 20 Gy
* Focuses of extra-hepatic liver uptake.
* Patients that cannot tolerate addition follow-up imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting with either primary or metastatic hepatic malignancies are the study population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Complications | 6 months
  Adverse Events related with the procedure
LPFS | 2 years
  Liver Progression Free Survival after the procedure
Tumor Response | 2 years
  Complete Response will be measured with the LI-RADS criteria for treatment response (LR-TR). In addition, RECIST v1.1, mRECIST, and PET-RECIST criteria will be further evaluated.

SECONDARY OUTCOMES:
Post-treatment dosimetry analysis | 2 years
  Correlate the safety and efficacy with the post-treatment dosimetry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Platon Dimopoulos, Resident, Study Director — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No